CLINICAL TRIAL: NCT04379466
Title: Effector and Regulatory T Cell Receptor Repertoire Analyses in Patients Affected by COVID-19
Acronym: CovRep
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200544; 2020-A01245-34 (Other: IDRCB)
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: COVID-19; T cell receptor; Effector T cells; Regulatory T cells; Single cell sequencing; Modelisation; Pathophysiology; Biomarkers
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The specificity of the adaptive immune response (AIR), and its balance between effector T cells (Teffs) and regulatory T cells (Tregs), is most likely a major determinant of the outcome of a Covid-19 infection.

We aim to analyze (i) the cellular components and (ii) the specificity of the AIR to COVID-19 in 60 patients with moderate and severe form of the disease. This should have important implications for (i) understanding the pathophysiology of the disease, (ii) discovering biomarkers of severity and (iii) designing treatments and vaccines.

DETAILED DESCRIPTION:
The quality of the adaptive immune response (AIR) to COVID-19 probably determines the course of the disease. Therefore, a comprehensive knowledge of the immune response to COVID-19 is required to better anticipate its outcome and identify vaccine targets. In particular, the quality of an AIR can be investigated by immunophenotyping (enumerating immune cells and assessing their fitness) and by analyzing the T cell receptor (TCR) repertoire.

The cellular components of the AIR will be analyzed by a deep immunophenotyping generating >800 measures assessing immune cells quantitatively and qualitatively (Pitoiset et al.,2018). Combined with supervised and unsupervised analyses, it has the power to detect subtle/hidden abnormalities.

The specificity will be analyzed by studying the global T cell receptor (TCR) repertoire of separated Tregs and Teffs from peripheral blood, as well as by single cell sequencing of cells from bronchoalveolar lavages.

These combined approaches should uncover parameters/abnormalities of the AIR linked to the infection severity and outcome, and lead to a better understanding of the nature of the Tregs and Teffs repertoires against COVID-19. This will have important implications for (i) understanding the pathophysiology of the disease, (ii) discovering biomarkers of severity and (iii) designing treatments and vaccines.

ELIGIBILITY:
Inclusion criteria :

* Age≥18 and ≤75 years
* Presenting a confirmed diagnosis of COVID-19 disease in accordance with WHO diagnostic criteria;
* Good venous capital ;
* Affiliation to a social security system;
* Having declared his/her non-opposition to participation in research (for patients hospitalized in intensive care units who are not able to communicate, the non-opposition of a trusted person will be sought.)

Exclusion criteria :

* Still under the exclusion period from another biomedical study
* Psychiatric illness or addiction that could interfere with the ability to comply with the requirements of the protocol or to give consent to participate in the study;
* Patient benefiting from a legal protection measure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or women, aged 18 to 75, infected with SARS-CoV-2 and admitted to the Pitié-Salpêtrière hospital for treatment
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
A list of COVID-19 specific TCR sequences | at day1

SECONDARY OUTCOMES:
One or more measures from peripheral blood immunophenotyping that is/are associated with COVID-19 outcome | at day1
Group of COVID-19 specific TCR sequences that is associated with COVID-19 outcome | at day1

CONTACTS AND LOCATIONS:
Overall Officials: David KLATZMANN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitie Salpétrère, Paris, France